CLINICAL TRIAL: NCT00886145
Title: Effect of Using Low-magnitude High Frequency Mechanical Stimulation of Bone in Persons With Subacute SCI
Brief Title: Effect of Vibration Therapy on Bone in Persons With Sub-acute Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William A. Bauman, M.D. (U.S. Federal Agency)
Collaborators: Kessler Foundation (Other)
Responsible Party: Sponsor-Investigator, William A. Bauman, M.D., Director, James J. Peters Veterans Affairs Medical Center
Organization: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B4162C-10
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Results first posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-02

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries; Mechanical Stimulation; Vibration Plate
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vibration and No Vibration (Other): Vibration: Right Leg and No Vibration: Left Leg.
  Interventions: Device: Vibration: Right Leg and No Vibration: Left Leg.

INTERVENTIONS:
Device: Vibration: Right Leg and No Vibration: Left Leg. — Vibration- right leg: The subjects will undergo a mechanical vibration intervention (Juvent Vibrating plate) in the seated position, with a load of 50lbs will be added to the right leg by using an extra wide strap equipped with bungee cords, 5 sessions a week, and each session lasting 20 minutes for a total of 6 month.
  No Vibration-left leg: At each vibration training session, the left leg will serve as a control with a load of 50lbs added to the left leg using an extra wide strap equipped with bungee cords, 5 sessions a week, and each session lasting 20 minutes for a total of 6 month.

SUMMARY:
The purpose of this research study is to determine the effect of mechanical vibrations on bones of persons with spinal cord injury.

DETAILED DESCRIPTION:
One of the major complications in persons with spinal cord injury (SCI) is marked bone loss because it greatly predisposes to skeletal fractures, even after minimal trauma. The use of low magnitude mechanical stimulation has been shown to be both safe and effective in improving bone mass and strength in animal studies. This modality has also been shown a beneficial effect in children with disability and in postmenopausal women. The investigators are interested in obtaining data to determine the possible benefits that mechanical intervention with vibratory stimulation may have on bone in individuals with subacute SCI (e.g., >1 month after injury but <1 year). Changes in bone density and mass of the leg and arm will be determined by dual energy X-ray absorptiometry (DXA); bone architecture of the distal leg and distal arm will be determined by peripheral quantitative computed tomography; circulating metabolic markers of bone will also be performed.

OBJECTIVES

In persons with subacute spinal cord injury:

1. To determine differences in bone mineral mass and parameters of bone structural integrity of the stimulated tibia versus the unstimulated tibia.
2. To determine changes in the metabolic markers of bone resorption and formation in persons with subacute spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Males;
2. Age 18-65;
3. Non-ambulatory SCI, with ASIA level A or B (ASIA A or B at the time of enrollment);
4. Neurological level of injury C3-T10;
5. Duration of injury >1 month after injury but <1 year; and 6.25(OH)D levels 30ng/ml (patients with values <30ng/ml will be supplemented with vitamin D to normalize values prior to study participation).

Exclusion Criteria:

1. Osteoporosis or low bone mass as determined by medical history or DXA at the baseline visit;
2. Pressure ulcer that may be exacerbated by the experimental procedure;
3. Fracture of the lower extremity within the past 5 years;
4. Active heterotopic ossification (HO);
5. History of metabolic bone disease;
6. Knee replacement(s);
7. Metal hardware in the lower extremities;
8. Bisphosphonate administration;
9. Severe underlying chronic illness (cardiac, pulmonary, gastrointestinal, etc.);
10. Renal disease (creatinine clearance < 40 mL/min);
11. 25(OH)D levels <30ng/ml;
12. Endocrine disorders known to be associated with osteoporosis (hyperthyroidism, hypercortisolism, and/or hypogonadism);
13. Alcoholism;
14. Seizure disorders;
15. History of kidney stones; and
16. Compliance 85% for every month up to the 4-month time-point

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-06; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Bauman, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Spinal Cord Damage Research Center — http://www.scirc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Vibration: Right Leg and No Vibration: Left Leg: The subjects will undergo vibration intervention in the seated position, 5 sessions a week, each session lasting 20 minutes for 6 months. All footwear will be removed, but they may wear socks or be barefoot. Only the right leg will be vibrated and the left leg will serve as a control. The frequency and force of the vibrations will be approximately 35 Hz and 0.3 g.
  In additional load of 50lbs will be added to both legs by using an extra wide strap equipped with bungee cords.
Period: Overall Study
Arm/Group | Vibration: Right Leg and No Vibration: Left Leg
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Vibration- Right Leg and No Vibration-left Leg: The subjects will undergo a mechanical vibration intervention (Juvent Vibrating plate) in the seated position, with a load of 50lbs will be added to the right leg by using an extra wide strap equipped with bungee cords, 5 sessions a week, and each session lasting 20 minutes for a total of 6 month.
  At each vibration training session, the left leg will serve as a control with a load of 50lbs added to the left leg using an extra wide strap equipped with bungee cords, 5 sessions a week, and each session lasting 20 minutes for a total of 6 month.
Arm/Group | Vibration- Right Leg and No Vibration-left Leg
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Volumetric Bone Mineral Density (vBMD) at 6-Months
Description: Volumetric Bone Mineral Density of the Right and Left Distal Tibia as Determined by Peripheral Quantitative Computed Tomography
Time Frame: The Percent Change in vBMD from Baseline to 6 months after Mechanical Stimulation Vibration Therapy
Measure: Number; unit: Percent Change
Groups:
- Vibration- Right Leg: Vibration- right leg: The subjects will undergo a mechanical vibration intervention (Juvent Vibrating plate) in the seated position, with a load of 50lbs will be added to the right leg by using an extra wide strap equipped with bungee cords, 5 sessions a week, and each session lasting 20 minutes for a total of 6 month.
- No Vibration- Left Leg: No Vibration-left leg: At each vibration training session, the left leg will serve as a control with a load of 50lbs added to the left leg using an extra wide strap equipped with bungee cords, 5 sessions a week, and each session lasting 20 minutes for a total of 6 month.
Arm/Group | Vibration- Right Leg | No Vibration- Left Leg
Number analyzed (Participants) | 1 | 1
Percent Change | -11 | -5.7

ADVERSE EVENTS:
Time Frame: 1.5 years
Groups:
- Vibration- Right Leg:: Vibration- right leg: The subjects will undergo a mechanical vibration intervention (Juvent Vibrating plate) in the seated position, with a load of 50lbs will be added to the right leg by using an extra wide strap equipped with bungee cords, 5 sessions a week, and each session lasting 20 minutes for a total of 6 month.
- No Vibration-left Leg:: No Vibration-left leg: At each vibration training session, the left leg will serve as a control with a load of 50lbs added to the left leg using an extra wide strap equipped with bungee cords, 5 sessions a week, and each session lasting 20 minutes for a total of 6 month.
Arm/Group | Vibration- Right Leg: | No Vibration-left Leg:
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vibration- Right Leg: (N=1) | No Vibration-left Leg: (N=1)
Autonomic Dysreflexia (Nervous system disorders) | 1 (1) | 1 (1) — Patient developed severe autonomic dysreflexia resulting from bowel impaction and was hospitalized. Symptoms of autonomic treated at the emergency room and condition completely resolved the following day when bowel impaction was corrected.

LIMITATIONS AND CAVEATS:
Subject recruitment was untenable due to the physiological and psychological healing necessary during the sub-acute phase of spinal cord injury.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes